CLINICAL TRIAL: NCT04321317
Title: Accuracy of Air Displacement Plethysmography Compare to Dual X-ray Absorptiometry (DXA) in Girls With Anorexia Nervosa
Brief Title: Validation of BodPod in Pediatric Anorexia Nervosa
Acronym: PADAAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 69HCL20_0120
Record Dates: First submitted 2020-03-23; First posted 2020-03-25 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Anorexia Nervosa
MeSH Terms: conditions — Anorexia Nervosa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Undernourished Patients (Other): All patients included will be included in the unique arm of the study
  Interventions: Other: Measure of body composition by Air Displacement Plethysmography (ADP)

INTERVENTIONS:
Other: Measure of body composition by Air Displacement Plethysmography (ADP) — Each patient included will have one measure of body composition by Air Displacement Plethysmography (ADP) during the initial consultation in the referent center for food disorders of Lyon and one year later.

SUMMARY:
Anorexia nervosa is a severe cause of undernutrition. It leads to a dramatic decrease of weight with an important modification of the body composition. During the renutrition phase, disharmonious body composition recovery is a relapse factor. Dual X-ray absorptiometry (DXA) is the gold standard to study body composition in children with anorexia nervosa. But, due to technical limits, DXA analysis needs to take in account a potential failure to thrive with an adjustment on height. Moreover DXA needs an irradiation which does not allow close repeat measurements. Since several years, a simple, non-invasive, non-irradiant method for measure of body composition has been developed in pediatrics: the air displacement plethysmography (ADP). Actually, only one device is available for this measurement: the BodPod®. However, feasibility and accuracy of ADP compare to DXA have not been evaluated in pediatric anorexia nervosa. The aim of this study is to compare the accuracy of BodPod® compare to DXA in girls with anorexia nervosa.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged between 8 and 18 years
* Female with a diagnosis of anorexia nervosa according to the DSM V classification, restrictive type or hyperphagic / purgative access type, evolving for less than 3 years.
* Female who received explanations adapted to their level of understanding for this study
* Female who expressed their consent to participate to this study
* Female whose parents or holders of parental authority have been informed and signed free and informed consent
* Female affiliated to a social security scheme

Exclusion Criteria:

* Patients with psychotic symptoms
* Patients with claustrophobia
* Patients with severe respiratory disease

Ages: 8 Years to 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 10 (Actual)
Dates: Start 2021-04-19 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Accuracy of Air Displacement Plethysmography (ADP) for body fat mass measurement | 1 year
  The accuracy of Air Displacement Plethysmography (ADP) will be compare to Dual X-ray Absorptiometry (DXA) according to the percentage of body fat mass measurement.
  The hypothesis will be validating if difference in percentage in body fat mass between ADP and DXA is below the 4%.
  The measurement will be done two times at 1 year interval

SECONDARY OUTCOMES:
Acceptability of Air Displacement Plethysmography (ADP) by the patient compared to Dual X-ray Absorptiometry (DXA) | 1 year
  The questionnaire includes 3 questions after the ADP using simple analog visual scales adapted to children comprehension.
  The measurement will be done two times at 1 year interval
Accuracy of Air Displacement Plethysmography (ADP) compare to Bio Electrical Impedance (BEI) | 1 year
  The difference between percentage of body fat mass will quantified between ADP and BEI.
  The measurement will be done two times at 1 year interval
Longitudinal evolution of the percentage of body fat mass | 1 year
  The evolution of the percentage of body fat mass will be evaluated after 1 year of evolution.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre REférent pour l'Anorexie et les Troubles du Comportement Alimentaire de Lyon (CREATyon) - Hôpital Neurologique Pierre Wertheimer - Hospices Civils de Lyon, Bron, France

IPD SHARING:
Plan to Share IPD: No